CLINICAL TRIAL: NCT07277751
Title: Investigating the Validity and Reliability of the L Test in Geriatric Individuals
Brief Title: Validity and Reliability of the L Test in Geriatric Individuals
Status: Active, not recruiting | Type: Observational
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Nail Abidin Yaraşır, Research Assistant, Hasan Kalyoncu University
Other Study IDs: HasanKU-FTR-NAY-01
Record Dates: First submitted 2025-11-29; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Geriatric Individuals; Geriatric
Keywords: Geriatric assessment; Aged

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Geriatric Individuals: ≥65 years Able to understand instructions Able to walk independently (with or without minimal assistive device) MMSE ≥24 (Mini Mental State Examination) No acute medical condition

SUMMARY:
Age-related declines in mobility, gait speed, balance, and functional independence are major determinants of morbidity and fall risk among older adults. Widely used functional mobility assessments-such as the Timed Up and Go Test (TUG) and the 10-Meter Walk Test (10MWT)-provide valuable information but do not fully capture the multidimensional motor tasks required in daily life, such as turning, directional changes, sit-to-stand transitions, and combined mobility tasks. The L Test, originally developed as an expanded form of TUG, includes turning, curved-path walking and a longer walking distance, and may therefore offer a more comprehensive assessment of functional mobility. Although previous studies have demonstrated high test-retest reliability and significant correlations with TUG in clinical populations such as Parkinson's disease and chronic conditions, evidence regarding the reliability and validity of the L Test in healthy geriatric individuals is lacking. This study aims to address this gap by evaluating the psychometric properties of the L Test in older adults.

Purpose: The purposes of the study are to: Evaluate the test-retest reliability of the L Test in geriatric individuals. Determine its concurrent validity by examining relationships with TUG and 10MWT. Calculate measurement error indices including Standard Error of Measurement (SEM) and Minimal Detectable Change (MDC).

Hypotheses H1: The L Test is a valid assessment tool for older adults. H2: The L Test demonstrates acceptable test-retest reliability (ICC ≥ 0.70). H3: The L Test shows a strong correlation with TUG (r ≥ 0.50). H4: The L Test shows a strong correlation with 10MWT (r ≥ 0.50).

Study Design: A cross-sectional methodological study with repeated measures (test-retest) one week apart.

Participants: Target population: Adults aged ≥65 years who can independently ambulate at least 10 meters.

Sample size: 58 participants based on power analysis; increased to 70 to compensate for potential attrition.

Sampling: Simple random sampling.

Inclusion Criteria:

≥65 years of age Mini-Mental State Examination ≥24 Able to walk 10 meters independently Voluntary participation

Exclusion Criteria:

Lower limb surgery within the past 6 months Diagnosed cardiovascular, neurological, or pulmonary disease Visual or auditory impairments affecting test safety

Procedures Participants will complete: L Test, Timed Up and Go Test (TUG), 10-Meter Walk Test (10MWT; normal and fast speed). One week later, all assessments will be repeated under the same conditions.

Outcome Measures: Primary: L Test time (seconds)

Secondary:TUG time, 10MWT time (normal and fast pace), SEM and MDC values. Pearson correlation with TUG and 10MWT

Statistical Analysis:

Test-retest reliability: ICC Concurrent validity: Pearson correlation coefficient Measurement error: SEM, MDC Significance level: p < 0.05

Ethical Considerations: All tests conducted by trained physiotherapists. Continuous supervision to minimize fall risk. Written informed consent obtained. Participants may withdraw at any time. Confidentiality ensured

Expected Outcomes: The study is expected to:

Provide normative data for the L Test in the geriatric population Demonstrate the test's psychometric robustness Support the clinical use of the L Test for functional mobility screening Contribute to physiotherapy and geriatric rehabilitation literature

DETAILED DESCRIPTION:
Background Functional mobility declines significantly with aging due to sarcopenia, reduced neuromuscular coordination, impaired balance, and slower gait speed. These changes contribute to increased fall risk, reduced independence, and diminished quality of life in older adults. Accurate assessment tools are essential for identifying early functional deterioration, planning individualized rehabilitation interventions, and monitoring clinical outcomes.

Commonly used functional tests such as the TUG and 10MWT measure important aspects of mobility; however, they do not fully represent the complexity of real-life movement patterns. Daily activities often require multidirectional walking, pivoting, turning, and completing longer paths that challenge balance and coordination.

The L Test is a modification of the TUG and incorporates: Sit-to-stand, straight walking, turning, extended pathway walking, returning and sitting. This structure more closely resembles real-world functional mobility demands. Previous studies in clinical groups, including Parkinson's disease and chronic obstructive pulmonary disease, have demonstrated strong reliability (ICC > 0.90) and significant correlations with TUG and gait speed tests. However, no studies have systematically examined the psychometric properties of the L Test among healthy older adults.

Given the progressive aging of the population and the increasing need for precise mobility assessments, establishing the reliability and validity of the L Test in geriatric individuals is clinically important.

Objectives: The primary objective is to determine the test-retest reliability of the L Test. Secondary objectives include: Determining concurrent validity against TUG and 10MWT Calculating measurement error (SEM, MDC) Contributing to clinical decision-making by identifying cutoff values for functional mobility.

Study Design and Setting: This is a single-center, observational methodological study conducted at: Hasan Kalyoncu University Medical Research and Application Center, Gaziantep, Türkiye.

Participants will be assessed twice at a one-week interval to evaluate test-retest reliability and measurement consistency.

Participants and Sample Size: A total of 70 participants will be recruited.

Inclusion Criteria

≥65 years Able to understand instructions Able to walk independently (with or without minimal assistive device) MMSE ≥24 No acute medical condition

Exclusion Criteria:

Lower-limb surgery within 6 months Diagnosed neurological or cardiopulmonary disease Visual or auditory impairments preventing safe assessment.

Study Procedures

1. Informed Consent and Baseline Assessments: Participants will receive verbal and written explanations about the study. After informed consent: Demographic data will be recorded.Height, weight, BMI, chronic diseases, use of assistive devices documented
2. Functional Tests:All tests will be administered by trained physiotherapists. L Test Procedure:Starting seated in a standard chair. Standing up upon instruction. Walking 3 m straight. Turning left and walking 7 m. Returning via the same route. Sitting down again. Total distance: 20 m. Time recorded using a stopwatch

TUG Test:Standing from a chair. Walking 3 m, turning, returning, and sitting. Time recorded.

10MWT: Walking a 14-m walkway (10-m timed zone). Three trials at normal and fast speed. Average used for analysis

3. Retesting: The full test battery will be repeated 1 week later under identical conditions.

Outcome Measures

Primary Outcome:

L Test completion time (seconds) Secondary Outcomes TUG time 10MWT time SEM MDC Correlation between L Test and other mobility tests.

Data Management and Analysis: Data will be stored securely with coded identifiers, complying with national data protection regulations.

Statistical Analysis Plan:

ICC (2,1) for test-retest reliability Pearson correlation for concurrent validity SEM = SD × √(1 - ICC) MDC = SEM × 1.96 × √2 Descriptive statistics for demographic variables p < 0.05 considered statistically significant

Ethics, Safety, and Monitoring:

Ethical approval has been obtained All procedures follow the Declaration of Helsinki Trained physiotherapists will supervise tests to prevent falls Participants may withdraw at any time Adverse events (if any) will be documented and reported

Expected Impact This study is expected to: Provide the first comprehensive psychometric evaluation of the L Test in healthy older adults. Offer clinicians a valid and reliable tool for mobility screening. Support risk stratification for falls and mobility limitations. Guide clinical decision-making in geriatric rehabilitation.

Dissemination Plan Results will be submitted to: Peer-reviewed journals, National and international physiotherapy and geriatric conferences. Participants may request a summary of the study results.

ELIGIBILITY:
Inclusion Criteria:

* ≥65 years
* Able to understand instructions
* Able to walk independently (with or without minimal assistive device)
* MMSE (Mini Mental State Examination) ≥24
* No acute medical condition

Exclusion Criteria:

* Lower-limb surgery within 6 months
* Diagnosed neurological or cardiopulmonary disease
* Visual or auditory impairments preventing safe assessment

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: As explained in the section on inclusion criteria: ≥65 years, able to understand instructions, able to walk independently (with or without minimal assistive device), MMSE (Mini Mental State Examination) ≥24, no acute medical condition
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2026-03-21 (Estimated); Study Completion 2026-04-21 (Estimated)

PRIMARY OUTCOMES:
L Test Procedure | one week
  Starting seated in a standard chair. Standing up upon instruction. Walking 3 m straight. Turning left and walking 7 m. Returning via the same route. Sitting down again. Total distance: 20 m. Time recorded using a stopwatch.
  The L-test has far less well-established normative data and validated cut-offs for older adults than TUG or gait speed. Several recent reviews note a lack of age-specific reference values or consensus study-based cut-off scores for older community-dwelling adults. Because of this limited evidence base, the L-test is useful for within-person change (reliability, MDC) but less suitable for population screening using a single universal cut-off.

SECONDARY OUTCOMES:
Time Up and Go (TUG) Test | one week
  Standing from a chair. Walking 3 m, turning, returning, and sitting. Time recorded.
  A frequently cited threshold for increased fall risk in community-dwelling older adults is ≈13.5 seconds. This value is often used as a screening cut-off for elevated fall risk.< 10-12 s: general indicator of normal to good functional mobility for many community-dwelling older adults (younger/healthier seniors often complete in 8-10 s).12-13.5 s: transitional zone - many studies treat this range as the threshold for increased fall risk or functional limitation. > 20 s (or substantially higher): often indicates significant mobility limitation, need for mobility aid and high fall/hospitalization risk (context dependent).
10 Metre Walking Test (10 MWT) | one week
  Walking a 14-m walkway (10-m timed zone). Three trials at normal and fast speed. Average used for analysis.
  < 0.8 m/s - commonly referenced threshold associated with increased health risk, reduced community ambulation and higher risk of adverse outcomes. < 0.7 m/s - associated in some reports with increased risk of hospitalization and dependency in older adults. 0.4-0.8 m/s - interpreted as limited community ambulation (below 0.4 m/s is usually household ambulation only). These bands are commonly used for functional classification. ≥ 1.0 m/s - often taken as the threshold associated with safe and independent community mobility and lower risk of adverse outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan Kalyoncu University Medical Research and Application Center, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data are not shared due to ethical principles. Should your work be published as a scientific paper, the data may be available from the relevant publication. Data may also be shared upon request for inclusion in a meta-analysis or systematic review study.